CLINICAL TRIAL: NCT06926426
Title: Efficacy of Oral Exercise Training in Oral Frailty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH111-REC3-070
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Elderly (People Aged 65 or More); Swallowing Training on Muscle Strength; Dysphagia
Keywords: Oral frailty; oral exercise training; ultrasound
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Training Intervention Group (Experimental): Oral function training (12-week program)
  Interventions: Behavioral: oral function training
- Usual Care Group (No Intervention): None (participants receive standard care only)

INTERVENTIONS:
Behavioral: oral function training — A 12-week program including oral muscle strengthening, pronunciation drills, and swallowing-related exercises designed to improve oral function in older adults.
  Arms: Oral Training Intervention Group

SUMMARY:
As the elderly grow older, the quality and function of skeletal muscle are affected. Sarcopenia is commonly seen in the elderly, due to the loss of skeletal muscle mass and function, often resulting in loss of activity and weight. Oral frailty refers to the status of oral function decline. Several studies indicate the relationship between sarcopenia and oral frailty, which is assumed to be the predictor of sarcopenia. Oral frailty may also progress to presbyphagia over time, causing higher risk of malnutrition, dehydration, pneumonia, and poor quality of life. In addition, recently, the use of ultrasound can measure the distance and speed of the hyoid bone displacement, thus more clearly assessing the swallowing function. The investigators aim to analyze whether oral exercise training can promote the oral and swallowing performance of the residents with oral frailty, and the feasibility of ultrasound as swallowing function evaluation.

The investigators' study will enroll participants from residential long-term care facilities according to the screening of oral frailty. The participants will be equally arranged to experimental and control groups. The intervention strategies will be given after institutional education training. Oral exercise training will be performed by facility's primary caregiver with professionals' remote supervision for 12 weeks. Evaluation tools include hand grip strength, 6-meter walking test, body composition analysis check (BIA), repeated saliva swallowing test, eating dysfunction scale (EAT-10), Functional Oral Intake Scale (FOIS), quality of life questionnaires, tongue muscle strength test and ultrasound swallowing function test.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Currently consuming food orally

Exclusion Criteria:

* Previously diagnosed with dysphagia
* Progressive central nervous system or motor disorders (e.g., dementia, Parkinson's disease)
* New-onset central nervous system disease within the past 6 months (e.g., stroke, traumatic brain injury)
* New-onset head and neck cancer within the past 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Hyoid Bone Displacement | Baseline and Week 12
  Change in hyoid bone displacement during swallowing assessed by ultrasound
Tongue pressure | At baseline and after 12 weeks of intervention
  Change in maximum anterior tongue pressure measured using the IOPI device

SECONDARY OUTCOMES:
Eating Assessment Tool-10 (EAT-10) Score | Baseline and after 12 weeks
  The Eating Assessment Tool-10 (EAT-10) is a self-administered symptom-specific outcome measure for dysphagia.
  Scoring Range: 0 to 40 Higher Scores: Indicate worse swallowing function and more severe symptoms
Handgrip Strength | Baseline and after 12 weeks
  Change in maximum grip strength measured by dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan